CLINICAL TRIAL: NCT03362125
Title: Bronchiolitis: Evaluation of Wang's Score as a Predictor of the Duration of Oxygen Therapy in Bronchiolitis
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC15_3022 BRONCHOLITE
Record Dates: First submitted 2017-11-15; First posted 2017-12-05 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-11

CONDITIONS: Bronchiolitis
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluation of Wang's score as a predictor of the duration of oxygen therapy in bronchiolitis

DETAILED DESCRIPTION:
Bronchiolitis is a viral disease of very variable evolution going from a simple outpatient treatment to the necessity of hospitalization in intensive care.

This epidemic disease is found all year round with a seasonal peak from mid-October to late winter.

The risk factors for progression to severe or prolonged bronchiolitis have been highlighted, but the duration of hospitalization is difficult to predict, which leads to organizational difficulties in the services and additional anxiety for the families.

The management of beds during winter epidemics can be a source of difficulties for hospitalization services, with the need to temporarily increase reception places or transfer children to other hospitals.

Oxygen rescue is the main factor limiting the discharge of the pediatric ward. This criterion seems to us more suitable than the total duration of hospitalization.

Indeed, other factors such as the family environment or food difficulties can delay the child's departure from the service. Their assessment seems to be more subjective, their assessment may vary from one doctor to another.

Better management of beds during winter epidemics could help to avoid changes in service during hospitalization, thus facilitating relationships between caregivers and families.

ELIGIBILITY:
Inclusion Criteria:

* Infants under 2 years
* Infants consulting at the emergency department of the University Hospital of Rennes for a first or second episode of bronchiolitis with criteria for hospitalization

Exclusion Criteria:

* Children transferred from another department such as pediatric intensive care unit
* Children for whom Wang's score could not be established
* Child over 2 years old at diagnosis
* Child with a 3rd episode of bronchiolitis or more.

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants less than 2 years old visiting the emergency department of the University Hospital of Rennes for a first or second episode of bronchiolitis with criteria for hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-02-15 (Actual); Study Completion 2016-02-15 (Actual)

PRIMARY OUTCOMES:
Relationship between the duration of oxygen therapy and Wang's score | through oxygen therapy completion an average of 82 hours
  Linear regression, to try to model the duration in hours of oxygen therapy according to Wang's score

SECONDARY OUTCOMES:
length of hospital stay | until the end of hospitalization an average of 10 days
  Relationship between length of hospital stay in hours and Wang's score
use of oxygen therapy | until the end of hospitalization an average of 10 days
  Relationship between use of oxygen therapy and Wang's score
transfer in intensive care | until the end of hospitalization an average of 10 days
  Relationship between secondary transfer in intensive care and Wang's score

CONTACTS AND LOCATIONS:
Overall Officials: Sylvaine Lefeuvre, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, France

IPD SHARING:
Plan to Share IPD: No